CLINICAL TRIAL: NCT02446470
Title: Sinus Tarsi Versus Extensile Lateral Approach for Open Reduction Internal Fixation of Intra-articular Calcaneus Fractures
Brief Title: Sinus Tarsi Versus Extensile Lateral Approach for Calcaneus Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-026
Record Dates: First submitted 2015-04-30; First posted 2015-05-18 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Intra-articular Fractures
Keywords: calcaneus; fracture fixation, internal
MeSH Terms: conditions — Intra-Articular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sinus Tarsi approach (Experimental): The Sinus Tarsi approach is the surgical approach for the incision.
  Interventions: Procedure: Sinus Tarsi approach
- Extensile Lateral approach (Active Comparator): The Extensile Lateral approach is the surgical approach for the incision.
  Interventions: Procedure: Extensile Lateral approach

INTERVENTIONS:
Procedure: Sinus Tarsi approach — A straight incision is made on the lateral side of the foot from the tip of the fibula to the base of the fourth metatarsal which centers the incision over the sinus tarsi. Then careful dissection is made through the subcutaneous tissues to prevent damage to the sural nerve, peroneal tendons, and extensor digitorum brevis (EDB). The origin of EDB is identified and the muscle is released distal enough to fully visualize the fracture and articular surface of the calcaneus. Following exposure of the fracture and articular surface of the calcaneus, open reduction and restoration of the articular surface of the calcaneus will be achieved followed by stable fracture fixation with plates and screws as dictated by the specific fracture pattern.
  Arms: Sinus Tarsi approach
Procedure: Extensile Lateral approach — An L-shaped incision overlying the lateral wall of the calcaneus will be made, followed by sharp dissection of soft tissues in line with the skin incision down to the periosteum. Effort will be made to identify and protect the sural nerve, as it commonly crosses the surgical field with this approach. The soft tissue flap is retracted as a single unit as subperiosteal dissection is performed. Following exposure of the lateral wall of the calcaneus, open reduction and restoration of the articular surface of the calcaneus will be achieved followed by stable fracture fixation with plates and screws as dictated by the specific fracture pattern.
  Arms: Extensile Lateral approach

SUMMARY:
This study is a prospective, randomized controlled trial comparing the sinus tarsi approach to the extensile lateral approach for surgical fixation of calcaneus fractures.

It is hypothesized that open reduction and internal fixation of intra-articular calcaneus fractures using a sinus tarsi approach will provide equivalent fracture reduction and stable fixation with significantly decreased wound complication rates in comparison to an extensile lateral approach.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients ≥ 18 years of age
* Closed intra-articular calcaneus fractures
* Undergoing surgical fixation (CPT code 28415)
* Ability to understand and agree to informed consent

Exclusion Criteria:

* Patients < 18 years of age
* Open fractures
* Dislocations that require open reduction
* Previous calcaneus abnormality or injury
* Unable to understand or agree to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Wound complication rate | approximately one year
  There is an expected wound complication rate of up to 30% with this type of fracture. The difference in wound complication rate between the two surgical approaches will be the primary outcome measure. Wound complications will be defined by the presence of superficial or deep infections, skin edge necrosis, and soft tissue sloughing.

SECONDARY OUTCOMES:
Fracture healing | approximately one year
  On radiographic and clinical exam
Rate of sural nerve injury | approximately one year
Rate of peroneal tendon injury | approximately one year
Change in operative time | one day
Rate of secondary surgery | approximately one year
Visual Analog Scale | approximately one year
  Pain Score
American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scale | approximately one year
  Functional Outcome Score
Foot Function Index | approximately one year
  Functional Outcome Score
Short-Form 36 (SF-36) Health Survey | approximately one year
  Functional Outcome Score

CONTACTS AND LOCATIONS:
Overall Officials: Jesse F Doty, MD, Principal Investigator — University of Tennessee College of Medicine Chattanooga/Erlanger Health System
Locations (1):
- Erlanger Health System, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No